CLINICAL TRIAL: NCT05964777
Title: Efficacy and Safety of rTMS-tACS Stimulation on Improving Cognitive Function in Bipolar Disorder: a Randomized, Double-blind, Sham Controlled Study
Brief Title: rTMS-tACS Stimulation on Improving Cognitive Function in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Head of Department of Psychaitry , First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT20230058C-R1
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Bipolar Disorder in Remission
Keywords: repetitive transcranial magnetic stimulation，Transcranial alternating current stimulation，diffusion tensor imaging，bipolar disorder
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation (Active Comparator): rTMS and tACS have a profound impact on cognitive impairment.,The damaged neural circuit of DLPFC-DACC may lead to impaired cognitive function in bipolar disorder.We used DTI imaging technology to calculate the stimulus site.Using high-frequency rTMS and high-precision tACS stimulation,thus affect the nerve ring pathway , thereby rapidly, effectively and safely improving cognitive impairment with bipolar disorder in remission.the subjects were subjected to rTMS for 20 minutes per day with the stimulation intensity of 10Hz and 100% of the motion threshold(MT),stimulation time of each sequence was 5 seconds, stimulation interval was 15 seconds, 3000 pulses per day for 15 days, and the total number of pulses was 45000.
  tACS has 5 high-precision targets, the total current is 2mA, and the stimulation frequency is 40hz. Under true stimulation, the current fade in and out time is 10 seconds, and the stimulation time is 30 minutes.
  Interventions: Device: Repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation
- Repetitive Transcranial magnetic stimulation and sham transcranial alternating current stimulation (Placebo Comparator): the subjects were subjected to rTMS for 20 minutes per day with the stimulation intensity of 10Hz and 100% of the motion threshold(MT),stimulation time of each sequence was 5 seconds, stimulation interval was 15 seconds, 3000 pulses per day for 15 days, and the total number of pulses was 45000.
  tACS has 5 high-precision targets, the total current is 2mA, and the stimulation frequency is 40hz. Under sham stimulation, the current fade in and out time is 10 seconds, the other 29 minutes and 40 seconds, no real current passes through.
  Interventions: Device: Repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation
- Sham repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation (Placebo Comparator): The stimulus intensity was 20% of MT in the ShamComparator arm, and the remaining parameters were the same as the Active Comparator arm.
  tACS has 5 high-precision targets, the total current is 2mA, and the stimulation frequency is 40hz. Under true stimulation, the current fade in and out time is 10 seconds, and the stimulation time is 30 minutes.
  Interventions: Device: Repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation

INTERVENTIONS:
Device: Repetitive Transcranial magnetic stimulation and transcranial alternating current stimulation — with the rapid development of neuroregulatory technology, rTMS and tACS have a profound impact on cognitive impairment. The damaged neural circuit of DLPFC-DACC may lead to impaired cognitive function in bipolar disorder.We used DTI imaging technology to calculate the DLPFC cortical region corresponding to the strongest point of dlpfc and DACC fiber connection as the stimulus site.Using high-frequency rTMS and high-precision tACS stimulation,thus affect the nerve ring pathway , thereby rapidly, effectively and safely improving cognitive impairment with bipolar disorder in remission.

SUMMARY:
Based on the individualized positioning technology of diffusion tensor imaging (DTI), the purpose of this study is to explore a new stimulation target and protocol for the treatment of bipolar disorder in remission through the repetitive transcranial magnetic stimulation(rTMS) and transcranial alternating current stimulation（tACS）under neuronavigation，verify whether there is abnormal functional connectivity and structural connections between the dorsolateral prefrontal cortex (dlpfc) and the dorsal anterior cingulate gyrus (dacc) related to cognitive impairment in bipolar disorder in remission, which will contribute to further understand the relevant neural pathway and mechanism.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 14-45 years old, regardless of gender] 2.Meet DSM-V diagnostic criteria for bipolar depressive in remission 3.Young Mania Rating Scale (YMRS) ≤ 6 points; 4.Hamilton Depression Scale(HAMD-17)≤7 points; 5.Cognitive deficit questionnaire PDQ≥17 points; 6.Han nationality, right-handed; 7.More than 9 years of education.

Exclusion Criteria:

1. History of severe somatic or brain organic diseases and craniocerebral trauma;
2. Abnormal brain structure or any MRI contraindications were found by magnetic resonance examination;
3. Those who do not cooperate or cannot effectively complete the experiment;
4. Drug, alcohol or other psychoactive substance abusers;
5. Pregnant, lactating or planned pregnancy;
6. ECT or rTMS or tACS treatment was performed within six months.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-04-04 (Estimated)

PRIMARY OUTCOMES:
thinc-it | 0,3week
  THINC-it test suites: Used primarily to assess cognitive dimensions such as executive function, learning and memory, attention, and processing speed in patients with BD. The assessment was conducted before and after treatment, and consisted of five main parts:Spotter,Symbol Check,Code Breaker,Trails test,PDQ-5-D

CONTACTS AND LOCATIONS:
Overall Officials: ShaoHua Hu, MD, Study Director — Zhejiang University; China Zhejiang, Study Director — The First Affiliated Hospital of Zhejiang University [Recruiting] Hangzhou, Zhejiang, China, 310000 Contact: ShaoHua Hu, MD 13957162903 dorhushaoh
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wang M, Zhou H, Zhang X, Chen Q, Tong Q, Han Q, Zhao X, Wang D, Lai J, He H, Zhang S, Hu S. Alleviating cognitive impairments in bipolar disorder with a novel DTI-guided multimodal neurostimulation protocol: a double-blind randomized controlled trial. BMC Med. 2025 Jun 4;23(1):334. doi: 10.1186/s12916-025-04174-z. PMID 40468342